# Exercise and Neuromodulation in Women with Fibromyalgia:

# **Neurophysiological Adaptations and Clinical Effects**

Unique Protocol Id: 33B2024

Date of Document: 14/10/2024

Sponsor: Universidad Andrés Bello

Principal Investigator: Edith Elgueta Cancino

# Study Protocol: Exercise and Neuromodulation in Women with Fibromyalgia: Neurophysiological Adaptations and Clinical Effects

#### INTRODUCTION

Fibromyalgia (FM) is the third most common musculoskeletal condition among unspecific chronic pain conditions with a prevalence of 2.7% worldwide<sup>1</sup> and a ratio female to male 3:1<sup>2</sup>. FM is characterized by three cardinal symptoms<sup>1</sup>: widespread pain (i.e. generalized head-to-toes <sup>1</sup> and neuropathic symptoms such as paraesthesia <sup>3</sup> <sup>4</sup>), fatigue (physical and mental) and sleep disorders (insomnia, frequent awakening, non-restoring sleep) <sup>15-7</sup>.

Several non-pharmacological treatments are available for managing FM symptoms such as (i) patient education, (ii) psychotherapy, (iii) neuromodulation (transcranial direct current stimulations: tDCS) and (iv) exercise <sup>1</sup>. The exercise has shown effective for reduce pain, fatigue and improves functionality in fibromyalgia<sup>8</sup>. The Ottawa expert panel recommends aerobic exercise as a treatment for individuals with fibromyalgia <sup>9</sup>. Similarly, the European League Against Rheumatism <sup>10</sup> exercise has strong recommendation as well; specifically, aerobic exercise has a moderate effect size to reduce pain and to improve physical function <sup>11</sup>. Bush et al. (2002) <sup>12</sup> was conducted to examine the effects of aerobic exercise training in FM, reporting reduction in pain levels (11.4%), pain pressure threshold (28.1%) and improves aerobic performance (17.1%) <sup>12</sup>. Despite the positive results of exercise interventions, the effect of moderate intensity exercise is small <sup>13</sup> and the adherence of these exercise programs is variable, with a treatment dropouts between 5%-34%<sup>14</sup>.

Among the strategies to enhance these metrics, various components of physical training have been analyzed, including frequency, duration, type of exercise, and intensity. Interesting, the intensity can play an important role in modulating pain and fatigue <sup>15</sup>. In healthy subjects, has been reported high-intensity interval training (HIIT) generates positive effects in the physical performance, such as increase in maximum strength, muscle power and lean mass <sup>16</sup>. HIIT can modulate the corticospinal excitability, generates exercise enjoyment and increases opioids release in comparison to moderate intensity continuous aerobic exercise <sup>17-19</sup>. These three components can play an important role in increasing exercise adherence. Regarding FM, there are two studies that have shown HIIT decrease pain, anxiety, depression and improves functional capacity, sleep quality and QoL<sup>15 20</sup>.

On the other hand, exercise has limitations such as muscle soreness and fatigue, which are described as common physiological effects of initial training in individuals who are deconditioned. Another alternative that has been shown to be effective for modulation of pain in FM, is neuromodulation through transcranial Direct Current Stimulation (tDCS). The tDCS has been shown to increase endogenous  $\mu$ -opioids release in chronic pain  $^{21}$  and in healthy subjects improves the muscle endurance  $^{22}$ . The exercise and tDCS have shown effectiveness in management on pain, fatigue, sleep, anxiety, depression, and quality of life  $^{15\,20\,23\text{-}26}$ . This suggests the tDCS effects are complementary to exercise  $^{23}$ . However, further research is needed to confirm these findings, due to the lack of evidence about combined effects of HIIT and tDCS in FM. We hypothesized HIIT + tDCS will be more effective in

the modulating on clinical and neurophysiological variables in comparison than HIIT + sham and HIIT alone.

#### **OBJECTIVES**

# Primary objective

The study aims to compare the effectiveness HIIT + tDCS, HIIT + sham tDCS and HIIT alone in reducing pain in women with FM.

# Secondary objective

- o To identify changes after training HIIT + tDCS, HIIT + sham tDCS and HIIT alone on pain, clinical and neurophysiological variables.
- To determine the association between pain, clinical and neurophysiological variables of HIIT + tDCS, HIIT + sham tDCS and HIIT alone.

#### MEHTODS AND ANALYSIS

#### Trial design

This protocol is reported following the Standard Protocol Items: Recommendations for Interventional Trials Guide<sup>27</sup>. This is a single centre, 3 arm factorial randomized clinical trial (RCT). The participants will be randomized by age and intensity of pain (moderate-severe) using a random blocked randomization sequence after pre intervention measurements. We will use a 1:1:1 allocation ratio to HIIT + tDCS, HIIT + sham tDCS and HIIT. Other investigator of staff will be carried out the randomization and sequentially numbered sealed envelopes process.

Only one investigator responsible for all assessments and training sessions will be blinded to tDCS intervention. The volunteers will not be blinded to tDCS.

## Study setting

This is a single site study. All procedures will be carried out at the Musculoskeletal Laboratory, Andrés Bello University.

# Eligibility criteria

*Inclusion criteria:* will include women between 18-65 years old with a diagnosis of Fibromyalgia by physician according to the criteria of the American College of Rheumatology (ACR) 2016. Stable medical treatment for symptoms for a least 4 weeks prior to participation, reported pain equal or higher than 4/10 on numeric rating pain scale (moderate or severe pain) for more than 3 months, body mass index (BMI) between 18.5 and 39.9 kg m<sup>-2</sup>, stable doses medication for ≥4 weeks, Central Sensitization inventory ≥40 points, controlled high blood pressure.

Exclusion criteria: Present pain unrelated to Fibromyalgia (isolated inflammatory joint, cancer, infectious, traumatic, localized neuropathic or degenerative joint pain), intense headache, cerebral surgery, seizure/epilepsy, cardiovascular, lung, metabolic (II diabetes mellitus), retinopathy or neurological diseases (i.e. stroke and traumatic brain injury antecedents), severe psychiatric disorders, medication contraindicated by TMS, have a cochlear-ferromagnetic and cardiac pacemaker, drugs and alcohol abuse. Are currently pregnant/breastfeeding, under physical therapy treatment or have participated in a designed

sports or exercise training in systematic programs previous 3 months. Are unable to speak or read Spanish fluently (inability to understand the pain scale and cooperate in testing).

#### **INTERVENTION**

Exercise

HIIT familiarization

The participants will perform a physical conditioning protocol that includes two weeks with three times per week <sup>28</sup> of HIIT 80%-95% of maximum heart rate (HR) <sup>20</sup> in the following way:

| TIME | INTERVAL | PASSIVE<br>RECOVERY | SESSIONS | maximum<br>HR |
|------|----------|---------------------|----------|---------------|
| 15 s | 2 | 2 min | 2 | 80%-95% |
| 30 s | 3-5 | 2 min | 2 | 80%-95% |
| 45 s | 5-7 | 2 min | 2 | 80%-95% |

Table 1. Description of HIIT familiarization.

#### HIIT training

From the seventh session to the eighteenth, the participants will perform a HIIT protocol that consists of 1 minute of active cycling at 80%-95% maximum HR  $^{20}$ , 2 minutes of passive recovery for 10 times (1x2x10). Moreover, during HIIT training, will be monitored the effort of HIIT session through RPE scale (6-20)  $^{29}$  at 15-18 RPE  $^{30 \ 31}$  between 50-60 revolutions per minute ("workload it costs to pedal, neither light nor heavy"), HR and pain at the beginning and end of each cycle of HIIT. If the participant fails to recover within 2 minutes (>70% maximum heart rate), longer rest time will be allowed until  $\leq$  70% of maximum HR is achieved  $^{28}$ . The maximum HR of each session will be considered the maximum HR for the HIIT prescription for the next session. In addition, the diet will be controlled with respect to the day before and the day of exercise session.

### Transcranial direct current stimulation (tDCS)

Over the course of four weeks, the tDCS will be applied at the same time as the HIIT session (during exercise). The individual will receive a total of 12 tDCS sessions.

#### Active (anodal) tDCS

The anode will be placed on the left M1 and the cathode on contralateral supraorbital area before the exercise starts. The stimulation will start at the same time the start exercise intervention, with an intensity of 2mA for 20 minutes <sup>32</sup>.

#### Sham tDCS

During exercise intervention, to replicate the feeling of current ramping up during active stimulation, the active anode placed on the left M1 will be activated for 30 seconds at the beginning and end of the procedure <sup>33</sup>. A period of 30 seconds of ramping is reliable for blinding <sup>34</sup>. Evidence shows that a time period of less than 3 minutes of tDCS intervention, does not generates cortical excitability changes <sup>33</sup>.

#### Outcomes

# Primary clinical outcome

The primary outcome is the Numeric rating scale (0-10). Commonly used to assess pain severity using a 0–10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable" <sup>35</sup>.

# Secondary clinical outcomes

The other cardinal symptoms in fibromyalgia are fatigue and sleep alterations. The fatigue will be assessed through the Multidimensional Fatigue Inventory (MFI)<sup>36</sup>. Sleep will be assessed through VAS (0-100mm)<sup>37</sup> and Pittsburgh Sleep Quality Index (PSQI)<sup>38</sup>.

Also, women with fibromyalgia suffer in psychosocial features and will be evaluated catastrophizing of pain through Pain Catastrophizing Scale (PCS)<sup>39</sup>, fear of movement through The Tampa Scale for Kinesiophobia (TSK)<sup>40-42</sup>, anxiety through State Trait Anxiety Inventory (STAI)<sup>43</sup> and depression through Beck's Depression Inventory II (BDI-II)<sup>44 45</sup>. The cardinal symptoms and psychosocial features affect the QoL. Will be evaluated the QoL through Fibromyalgia Impact Questionnaire (FIQ)<sup>46</sup> and Short Form 36<sup>47</sup>.

Regarding exercise, will be evaluated the Three-repetition sit-to-stand test (3R-STS) to quantify the muscle soreness before training sessions, the individuals will be asked to sit and stand 3 times with their legs shoulder width apart and bend their knees to 90° <sup>48</sup> by the VAS pain (0-100 mm). The VAS pain is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain" <sup>49</sup>. The volunteers must mark with a straight vertical line on the horizontal line. Moreover, will be assessed exercise adherence through Exercise Attitude Questionnaire-18 (EAQ-18) <sup>50</sup> <sup>51</sup>, exercise enjoyment through Physical Activity Enjoyment Scale (PACES)<sup>52</sup> <sup>53</sup>, physical level activity through International Physical Activity Questionnaire (IPAQ)<sup>54</sup> and cardiovascular risk through Physical Activity Readiness Questionnaire (PAR-Q)<sup>55</sup>, the perception of effort during the exercise by Borg's Scale <sup>56</sup> and dyspnoea<sup>57</sup> <sup>58</sup>. Finally, will be assessed the anthropometric characteristics through InBody 770 (Sout Korea) and the heigh by stadiometer.

## Secondary neuro-physiological outcomes

The corticospinal excitability will be measured with transcranial magnetic stimulation using a Magstim 200<sup>2</sup> & a 7 mm double cone coil (Magstim, UK) in combination with surface electromyography (sEMG; Delsys Bagnoli 16 channels, USA) (supplementary information 10). The stimulation will be in left M1 cortex, and the EMG recordings will be gathered in right vastus lateralis muscle using Ag/AgCl electrodes. The specific variables that will be assessed are:

Motor Evoked Potential (MEP): is the response of the muscle to the stimulation of the corticomotor pathway and it is frequently used to estimate corticospinal excitability <sup>59</sup>. It can be measured as the peak-to-peak amplitude of the EMGs signal. The average of 15 MEPs peak-to-peak amplitudes using an intensity of 120% active motor threshold (aMT) will be collected to asses CSE <sup>60 61</sup>.

Cortical Silent Period (CSP): The CSP is defined as the "temporary interruption of electromyographic signal from muscle following a MEP" <sup>62</sup>. It is considered a measure of the excitability mediated by gamma-aminobutyric acid (GABA<sub>B</sub>) receptors (GABA<sub>B</sub>R). The SP will be measured in milliseconds (ms) from the end of the MEP wave to the recovery EMG signal to the basal averaged amplitud <sup>63</sup> <sup>64</sup>.

Rest Motor Threshold (rMT, % output): rMT is defined as the lowest stimulus intensity to evoke MEPs with a peak-to-peak amplitude of  $50\mu V$  in at least five out of 10 consecutive trials when the muscle at rest  $^{65}$ . rMT will be expressed as percentage of the TMS output.

Active Motor Threshold (aMT, % output): it is the lowest intensity of the stimulator needed to evoke MEPs with a peak-to-peak amplitude of  $\geq 200 \,\mu\text{V}$  in five out of 10 consecutive trials while maintaining an isometric contraction at 10% of the maximal voluntary contraction (MVC)<sup>66</sup>. aMT will be expressed as percentage of the TMS output.

Short Interval intracortical Inhibition (SICI) and Intracortical Facilitation (ICF): Both are transient phenomena that occur at the motor cortex, SICI is a suppression or reduction of the firing of cortical neurons - GABA<sub>A</sub> inhibitory circuits- <sup>67-69</sup> and ICF is an excitatory phenomenon mediated by N-methyl-D-aspartate receptors (NMDAR) <sup>70</sup>. Paired pulse paradigms will be used to assess both. These paradigms involve two consecutive stimulations, one conditioning stimulus that is below the threshold (80% rMT) followed by a test stimulus that is above the threshold (120% of the motor threshold) <sup>32</sup>. To assess short intracortical inhibition (SICI), the interstimulus interval will be set to 2 ms, while for intracortical facilitation (ICF), the interval will be set to 15 ms <sup>32</sup>. We will administer ten random stimuli at each interval and calculate the percentage of inhibition or facilitation before and after treatment <sup>32</sup>.

Others neuro-physiological outcomes will be assessed are pain pressure threshold by algometer in bilateral supraspinatus muscle, lateral epicondyle, gluteus area and medial fat knee according ACR 1990 <sup>71 72</sup>, aerobic capacity <sup>73</sup>, quadriceps strength of dominant leg by maximal voluntary isometric contraction (MVIC) <sup>74</sup> and endurance muscle contraction by a time to exhaustion of knee extensors (20% MVIC) adding to High density electromyography (HD-sEMG) for motor units recruitment <sup>75-77</sup>.

#### STATISTICAL ANALYSIS PLAN

#### Study sample

Will include women between 18-65 years old with a diagnosis of Fibromyalgia by physician according to the criteria of the American College of Rheumatology (ACR) 2016. We will enroll 40 volunteers divided into 3 groups.

# Sample size calculation

The sample size was calculated using G\*Power 3.1 (Germany), based on the variable pain measured by the Visual Analogue Scale (VAS) from the study by Kolak et al.  $(2022)^{78}$  with a power of 0.80, an alpha level of 0.05, and accounting for a 20% dropout rate, the required sample size was determined a total of n=40.

#### Statistical Analysis

The distribution of the data for all variables will be corroborated with the Shapiro wilk normality test. Two-way ANOVA and Pearson correlation will be used if the data is normally distributed, considering a p value < 0.05. If no normal distribution is found the data will be transformed or nonparametric analysis will be used. The data will be presented as mean and standard deviation. Moreover, Two-way ANCOVA will be performed.

# Ethics and dissemination

This protocol was approved by the scientific ethics committee (number: 33B2024) at the Faculty of Medicine, Andres Bello University. The results will be reported in congress and peer review journal.

#### REFERENCES

- 1. Sarzi-Puttini P, Giorgi V, Marotto D, et al. Fibromyalgia: an update on clinical characteristics, aetiopathogenesis and treatment. *Nat Rev Rheumatol* 2020;16(11):645-60. doi: 10.1038/s41584-020-00506-w [published Online First: 2020/10/08]
- 2. Queiroz LP. Worldwide epidemiology of fibromyalgia. *Current pain and headache reports* 2013;17:1-6.
- 3. Koroschetz J, Rehm SE, Gockel U, et al. Fibromyalgia and neuropathic pain-differences and similarities. A comparison of 3057 patients with diabetic painful neuropathy and fibromyalgia. *BMC neurology* 2011;11(1):1-8.
- 4. Rehm SE, Koroschetz J, Gockel U, et al. A cross-sectional survey of 3035 patients with fibromyalgia: subgroups of patients with typical comorbidities and sensory symptom profiles. *Rheumatology* 2010;49(6):1146-52.
- 5. Sandıkçı SC, Özbalkan Z. Fatigue in rheumatic diseases. *European Journal of Rheumatology* 2015;2(3):109.
- 6. Kleinman L, Mannix S, Arnold LM, et al. Assessment of sleep in patients with fibromyalgia: qualitative development of the fibromyalgia sleep diary. *Health and quality of life outcomes* 2014;12:1-11.
- 7. Bennett RM, Jones J, Turk DC, et al. An internet survey of 2,596 people with fibromyalgia. *BMC musculoskeletal disorders* 2007;8(1):1-11.
- 8. Geneen LJ, Moore RA, Clarke C, et al. Physical activity and exercise for chronic pain in adults: an overview of Cochrane Reviews. *Cochrane Database Syst Rev* 2017;4(4):CD011279. doi: 10.1002/14651858.CD011279.pub3 [published Online First: 2017/04/25]
- 9. Brosseau L, Wells GA, Tugwell P, et al. Ottawa Panel evidence-based clinical practice guidelines for aerobic fitness exercises in the management of fibromyalgia: part 1. *Phys Ther* 2008;88(7):857-71. doi: 10.2522/ptj.20070200 [published Online First: 2008/05/24]
- 10. Macfarlane GJ, Kronisch C, Dean LE, et al. EULAR revised recommendations for the management of fibromyalgia. *Ann Rheum Dis* 2017;76(2):318-28. doi: 10.1136/annrheumdis-2016-209724 [published Online First: 2016/07/06]
- 11. Busch AJ, Barber KA, Overend TJ, et al. Exercise for treating fibromyalgia syndrome. *Cochrane database of systematic reviews* 2008(4)
- 12. Busch A, Schachter CL, Peloso PM, et al. Exercise for treating fibromyalgia syndrome. *Cochrane Database Syst Rev* 2002(3):CD003786. doi: 10.1002/14651858.CD003786 [published Online First: 2002/07/26]
- 13. Hauser W, Klose P, Langhorst J, et al. Efficacy of different types of aerobic exercise in fibromyalgia syndrome: a systematic review and meta-analysis of randomised controlled trials. *Arthritis Res Ther* 2010;12(3):R79. doi: 10.1186/ar3002 [published Online First: 2010/05/13]
- 14. Sarmento CV, Liu Z, Smirnova IV, et al. Exploring Adherence to Moderate to High-Intensity Exercises in Patients with Fibromyalgia: The Role of Physiological and Psychological Factors—A Narrative Literature Review. *Physiologia* 2023;3(3):472-83.
- 15. Bodéré C, Cabon M, Woda A, et al. A training program for fibromyalgia management: A 5-year pilot study. *SAGE Open Medicine* 2020;8:2050312120943072.

- 16. Caparrós-Manosalva C, Garrido-Muñoz N, Alvear-Constanzo B, et al. Effects of highintensity interval training on lean mass, strength, and power of the lower limbs in healthy old and young people. *Frontiers in Physiology* 2023;14
- 17. Saanijoki T, Tuominen L, Tuulari JJ, et al. Opioid release after high-intensity interval training in healthy human subjects. *Neuropsychopharmacology* 2018;43(2):246-54.
- 18. Thum JS, Parsons G, Whittle T, et al. High-intensity interval training elicits higher enjoyment than moderate intensity continuous exercise. *PloS one* 2017;12(1):e0166299.
- 19. Hendy AM, Andrushko JW, Della Gatta PA, et al. Acute effects of high-intensity aerobic exercise on motor cortical excitability and inhibition in sedentary adults. *Frontiers in Psychology* 2022;13:814633.
- 20. Atan T, Karavelioğlu Y. Effectiveness of high-intensity interval training vs moderate-intensity continuous training in patients with fibromyalgia: a pilot randomized controlled trial. *Archives of Physical Medicine and Rehabilitation* 2020;101(11):1865-76.
- 21. DosSantos MF, Love TM, Martikainen IK, et al. Immediate effects of tDCS on the μ-opioid system of a chronic pain patient. *Frontiers in psychiatry* 2012;3:93.
- 22. Cogiamanian F, Marceglia S, Ardolino G, et al. Improved isometric force endurance after transcranial direct current stimulation over the human motor cortical areas. *European Journal of Neuroscience* 2007;26(1):242-49.
- 23. Mendonca ME, Simis M, Grecco LC, et al. Transcranial direct current stimulation combined with aerobic exercise to optimize analgesic responses in fibromyalgia: a randomized placebo-controlled clinical trial. *Frontiers in human neuroscience* 2016;10:68.
- 24. Teixeira PE, Pacheco-Barrios K, Branco LC, et al. The analgesic effect of transcranial direct current stimulation in fibromyalgia: a systematic review, meta-analysis, and meta-regression of potential influencers of clinical effect. *Neuromodulation: Technology at the Neural Interface* 2023;26(4):715-27.
- 25. Hou W-H, Wang T-Y, Kang J-H. The effects of add-on non-invasive brain stimulation in fibromyalgia: a meta-analysis and meta-regression of randomized controlled trials. *Rheumatology* 2016;55(8):1507-17.
- 26. Couto N, Monteiro D, Cid L, et al. Effect of different types of exercise in adult subjects with fibromyalgia: a systematic review and meta-analysis of randomised clinical trials. *Scientific Reports* 2022;12(1):10391.
- 27. Chan A-W, Tetzlaff JM, Gøtzsche PC, et al. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. *Bmj* 2013;346
- 28. Cano-Montoya J, Álvarez C, Martínez C, et al. Recuperación cardiovascular durante ejercicio intermitente en pacientes con hipertensión y diabetes tipo 2 altamente adherentes. *Revista médica de Chile* 2016;144(9):1150-58.
- 29. Abbiss CR, Peiffer JJ, Meeusen R, et al. Role of ratings of perceived exertion during self-paced exercise: what are we actually measuring? *Sports medicine* 2015;45:1235-43.
- 30. Taylor JL, Holland DJ, Spathis JG, et al. Guidelines for the delivery and monitoring of high intensity interval training in clinical populations. *Progress in cardiovascular diseases* 2019;62(2):140-46.
- 31. Taylor JL, Bonikowske AR, Olson TP. Optimizing outcomes in cardiac rehabilitation: the importance of exercise intensity. *Frontiers in Cardiovascular Medicine* 2021;8:734278.

- 32. Castelo-Branco L, Kucukseymen EU, Duarte D, et al. Optimised transcranial direct current stimulation (tDCS) for fibromyalgia—targeting the endogenous pain control system: a randomised, double-blind, factorial clinical trial protocol. *BMJ open* 2019;9(10)
- 33. Nitsche MA, Paulus W. Excitability changes induced in the human motor cortex by weak transcranial direct current stimulation. *The Journal of physiology* 2000;527(Pt 3):633.
- 34. Gandiga PC, Hummel FC, Cohen LG. Transcranial DC stimulation (tDCS): a tool for double-blind sham-controlled clinical studies in brain stimulation. *Clinical neurophysiology* 2006;117(4):845-50.
- 35. Breivik H, Pc B. Allen sm, et al. Assessment of pain Br J Anaesth 2008;101:17-24.
- 36. Munguía-Izquierdo D, Segura-Jiménez V, Camiletti-Moirón D, et al. Multidimensional Fatigue Inventory: Spanish adaptation and psychometric properties for fibromyalgia patients. The Al-Andalus study. *Clin Exp Rheumatol* 2012;30(Suppl 74):94-102.
- 37. Martin S, Chandran A, Zografos L, et al. Evaluation of the impact of fibromyalgia on patients' sleep and the content validity of two sleep scales. *Health and Quality of Life Outcomes* 2009;7:1-7.
- 38. Hita-Contreras F, Martínez-López E, Latorre-Román PA, et al. Reliability and validity of the Spanish version of the Pittsburgh Sleep Quality Index (PSQI) in patients with fibromyalgia. *Rheumatology international* 2014;34:929-36.
- 39. Campayo JG, Rodero B, Alda M, et al. Validación de la versión española de la escala de la catastrofización ante el dolor (Pain Catastrophizing Scale) en la fibromialgia. *Medicina Clinica* 2008;131(13):487-92.
- 40. Roelofs J, Goubert L, Peters ML, et al. The Tampa Scale for Kinesiophobia: further examination of psychometric properties in patients with chronic low back pain and fibromyalgia. *European Journal of Pain* 2004;8(5):495-502.
- 41. Burwinkle T, Robinson JP, Turk DC. Fear of movement: factor structure of the Tampa Scale of Kinesiophobia in patients with fibromyalgia syndrome. *The Journal of pain* 2005;6(6):384-91.
- 42. Gómez-Pérez L, López-Martínez AE, Ruiz-Párraga GT. Psychometric properties of the Spanish version of the Tampa Scale for Kinesiophobia (TSK). *The journal of Pain* 2011;12(4):425-35.
- 43. Spielberger CD, Gorsuch RL, Lushene RE. Cuestionario de ansiedad estado-rasgo. *Madrid: Tea* 1982;1
- 44. Sanz J, Perdigón A, Vázquez C. The Spanish adaptation of Beck's Depression Inventory-II (BDI-II): 2. Psychometric properties in the general population. *Clínica y Salud* 2003;14(3):249-80.
- 45. Beck AT, Steer RA, Brown G. Beck depression inventory–II. *Psychological assessment* 1996
- 46. Salgueiro M, García-Leiva JM, Ballesteros J, et al. Validation of a Spanish version of the revised fibromyalgia impact questionnaire (FIQR). *Health and quality of life outcomes* 2013;11(1):1-8.
- 47. Monterde S, Salvat I, Montull S, et al. Validación de la versión española del Fibromyalgia Impact Questionnaire. *Rev esp reumatol(Ed impr)* 2004:507-13.
- 48. Aldayel A, Jubeau M, McGuigan MR, et al. Less indication of muscle damage in the second than initial electrical muscle stimulation bout consisting of isometric contractions of the knee extensors. *European journal of applied physiology* 2010;108:709-17.

- 49. Delgado DA, Lambert BS, Boutris N, et al. Validation of digital visual analog scale pain scoring with a traditional paper-based visual analog scale in adults. *Journal of the American Academy of Orthopaedic Surgeons Global research & reviews* 2018;2(3)
- 50. Arturi P, Schneeberger EE, Sommerfleck F, et al. Adherence to treatment in patients with ankylosing spondylitis. *Clinical rheumatology* 2013;32:1007-15.
- 51. Manigandan C, Charles J, Divya I, et al. Construction of exercise attitude questionnaire-18 to evaluate patients' attitudes toward exercises. *International Journal of Rehabilitation Research* 2004;27(3):229-31.
- 52. Motl RW, Dishman RK, Saunders R, et al. Measuring enjoyment of physical activity in adolescent girls. *American journal of preventive medicine* 2001;21(2):110-17.
- 53. Moreno J-A, González-Cutre D, Martínez C, et al. Propiedades psicométricas de la Physical Activity Enjoyment Scale (PACES) en el contexto español. *Estudios de Psicología* 2008;29(2):173-80.
- 54. Craig CL, Marshall AL, Sjöström M, et al. International physical activity questionnaire: 12-country reliability and validity. *Medicine & science in sports & exercise* 2003;35(8):1381-95.
- 55. Baechle TR, Earle R, Baechle TR. NSCA's essentials of personal training: Human Kinetics 2004.
- 56. Borg G. Borg's perceived exertion and pain scales: Human kinetics 1998.
- 57. Crisafulli E, Clini EM. Measures of dyspnea in pulmonary rehabilitation. *Multidisciplinary respiratory medicine* 2010;5:1-9.
- 58. Inostroza M, Valdés O, Tapia G, et al. Effects of eccentric vs concentric cycling training on patients with moderate COPD. *European journal of applied physiology* 2022:1-14.
- 59. Klomjai W, Katz R, Lackmy-Vallee A. Basic principles of transcranial magnetic stimulation (TMS) and repetitive TMS (rTMS). *Ann Phys Rehabil Med* 2015;58(4):208-13. doi: 10.1016/j.rehab.2015.05.005 [published Online First: 2015/09/01]
- 60. Ridding M, Taylor J. Mechanisms of motor-evoked potential facilitation following prolonged dual peripheral and central stimulation in humans. *The Journal of physiology* 2001;537(2):623-31.
- 61. Bement MKH, Weyer AD, Yoon T, et al. Corticomotor excitability during a noxious stimulus before and after exercise in women with fibromyalgia. *Journal of Clinical Neurophysiology* 2014;31(1):94-98.
- 62. Zeugin D, Ionta S. Anatomo-functional origins of the cortical silent period: spotlight on the basal ganglia. *Brain sciences* 2021;11(6):705.
- 63. Hupfeld K, Swanson C, Fling B, et al. TMS-induced silent periods: A review of methods and call for consistency. *Journal of neuroscience methods* 2020;346:108950.
- 64. Cacchio A, Cimini N, Alosi P, et al. Reliability of transcranial magnetic stimulation-related measurements of tibialis anterior muscle in healthy subjects. *Clinical neurophysiology* 2009;120(2):414-19.
- 65. Pacheco-Barrios K, Lima D, Pimenta D, et al. Motor cortex inhibition as a fibromyalgia biomarker: A meta-analysis of transcranial magnetic stimulation studies. *Brain network and modulation* 2022;1(2):88.
- 66. Groppa S, Oliviero A, Eisen A, et al. A practical guide to diagnostic transcranial magnetic stimulation: report of an IFCN committee. *Clin Neurophysiol* 2012;123(5):858-82. doi: 10.1016/j.clinph.2012.01.010 [published Online First: 2012/02/22]

- 67. Kujirai T, Caramia M, Rothwell JC, et al. Corticocortical inhibition in human motor cortex. *The Journal of physiology* 1993;471(1):501-19.
- 68. Ziemann U, Lönnecker S, Steinhoff B, et al. Effects of antiepileptic drugs on motor cortex excitability in humans: a transcranial magnetic stimulation study. *Annals of Neurology: Official Journal of the American Neurological Association and the Child Neurology Society* 1996;40(3):367-78.
- 69. Ziemann U, Rothwell JC, Ridding M. Interaction between intracortical inhibition and facilitation in human motor cortex. *The Journal of physiology* 1996;496(3):873-81.
- 70. Wagle-Shukla A, Ni Z, Gunraj CA, et al. Effects of short interval intracortical inhibition and intracortical facilitation on short interval intracortical facilitation in human primary motor cortex. *The Journal of physiology* 2009;587(23):5665-78.
- 71. Kosek E, Ekholm Ja, Nordemar R. A comparison of pressure pain thresholds in different tissues and body regions. Long-term reliability of pressure algometry in healthy volunteers. *Scandinavian journal of rehabilitation medicine* 1993;25(3):117-24.
- 72. Wolfe F, Smythe HA, Yunus MB, et al. The American College of Rheumatology 1990 criteria for the classification of fibromyalgia. *Arthritis & Rheumatism: Official Journal of the American College of Rheumatology* 1990;33(2):160-72.
- 73. Hooten WM, Smith JM, Eldrige JS, et al. Pain severity is associated with muscle strength and peak oxygen uptake in adults with fibromyalgia. *Journal of pain research* 2014:237-42.
- 74. Martinez-Valdes E, Falla D, Negro F, et al. Differential motor unit changes after endurance or high-intensity interval training. *Med Sci Sports Exerc* 2017;49(6):1126-36.
- 75. Angius L, Pageaux B, Hopker J, et al. Transcranial direct current stimulation improves isometric time to exhaustion of the knee extensors. *Neuroscience* 2016;339:363-75.
- 76. Bouillard K, Jubeau M, Nordez A, et al. Effect of vastus lateralis fatigue on load sharing between quadriceps femoris muscles during isometric knee extensions. *Journal of neurophysiology* 2014;111(4):768-76.
- 77. Martinez-Valdes E, Laine C, Falla D, et al. High-density surface electromyography provides reliable estimates of motor unit behavior. *Clinical Neurophysiology* 2016;127(6):2534-41.
- 78. Kolak E, Ardıç F, Fındıkoğlu G. Effects of different types of exercises on pain, quality of life, depression, and body composition in women with fibromyalgia: A three-arm, parallel-group, randomized trial. *Archives of Rheumatology* 2022;37(3):444.